CLINICAL TRIAL: NCT00557843
Title: Influence of Continuous Bupivacaine Infusion on Tissue Oxygenation Following Colonic Surgery
Brief Title: Continuous Bupivacaine Infusion Following Colonic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 07-758
Record Dates: First submitted 2007-11-13; First posted 2007-11-14 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2017-04

CONDITIONS: Abdominal Surgery
Keywords: Bupivacaine; Colon; Surgery; Oxygenation
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- bupivacaine (Active Comparator): Wound perfusion with bupivacaine, plus patient controlled analgesia (PCA)
  Interventions: Drug: Bupivacaine
- Placebo (Placebo Comparator): Wound perfusion with placebo solution (isotonic saline) plus patient controlled analgesia (PCA)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Bupivacaine — Wound perfusion with bupivacaine, plus patient controlled analgesia (PCA)
  Other Names: Marcain, Marcaine,Sensorcaine
  Arms: bupivacaine
Drug: Saline — Wound perfusion with placebo solution (isotonic saline) plus patient controlled analgesia (PCA)
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate the influence of continuous local anesthetic infiltration on tissue oxygenation after surgical procedures requiring abdominal surgery as a major predictor for wound healing.

DETAILED DESCRIPTION:
Patients undergoing abdominal surgery will be randomized to one of two groups.

Group 1: Wound perfusion with bupivacaine, plus patient controlled analgesia (PCA)

Group 2: Wound perfusion with placebo solution (isotonic saline) plus patient controlled analgesia (PCA)

All patients will be premedicated with IV midazolam up to 5 mg. On arrival to the operating room, a fluid bolus of 10 ml/kg/h will be administered before induction of anesthesia.

Those randomized to local wound perfusion will receive the local anesthetic or placebo via the ON-Q pain management system. At the end of surgery a catheter will be positioned in the subcutaneous layer of the wound, leaving via a separate stab incision. The wound closure will then be completed.

A loading dose of local anesthetic solution, 20 ml lidocaine 1% plus 20 ml bupivacaine 0.5%, or, the same amount of placebo will be injected into the wound before the patient leaves the operating room. Thereafter bupivacaine 0.5% alone or placebo will be injected continuously into the wound at a flow rate of 2 ml/h for 24 hours.

Subcutaneous oxygen tension (PsqO2) will be evaluated intraoperatively with a polygraphic-type tissue oxygen sensor positioned within a subcutaneous, saline filled Silastic® tonometer inserted into the patients' upper arm after induction of anesthesia.

Postoperative pain relief will be maintained by patient-controlled analgesia (PCA) with morphine (2mg bolus, 6-minute lock-out) and with local anesthetic wound perfusion.

Patients will be given supplemental oxygen via a face mask at a rate of 2 L/min. Additional oxygen will be given as necessary to maintain an oxygen saturation > 95%.

An observer blinded to group assignment will perform all the postoperative evaluations.

Patient chart review will be undertaken to screen for evidence of surgical wound infection. The presence of infection will be determined by review of the attending surgeon's documentation in the patient's chart.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years of age.
2. The patient has provided written informed consent.
3. The patient is scheduled for abdominal surgery.
4. The patient has an ASA of I, II, or III.
5. The patient understands the explanation of the protocol.

Exclusion Criteria:

1. Patients aged < 18 and > 80 years.
2. History of diabetes mellitus.
3. History of congestive heart failure.
4. History of peripheral vascular disease.
5. History of smoking.
6. History of Dysautonomia.
7. History of thyroid disease.
8. Susceptibility to malignant hyperthermia.
9. History of morbid obesity.
10. History of fever
11. History of infection.
12. Contraindication to the placement of an arterial line; e.g., Raynaud's disease.
13. The patient declines participation.
14. Any patient the investigator feels is not a candidate for this study.
15. Any patient with a history of known alcohol, analgesic, or narcotic substance abuse within two years of screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
tissue oxygenation | 24 hours post surgery
  averge tissue oxygenation on wound healing after abdominal surgery

SECONDARY OUTCOMES:
Verbal rating scales (VRS) | 24 hours post surgery
  0 -10 scale with 0 = no pain and 10 = worst pain

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Kurz, MD, Principal Investigator — The Cleveland Clinic; Daniel I Sessler, MD, Study Chair — The Cleveland Clinic

IPD SHARING:
Plan to Share IPD: No